CLINICAL TRIAL: NCT01500200
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate ALKS 5461 in Subjects With Major Depressive Disorder and Inadequate Response to Antidepressant Therapy
Brief Title: A Study to Evaluate ALKS 5461 in Subjects With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK5461-202
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — ALKS 5461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALKS 5461 (Experimental)
  Interventions: Drug: ALKS 5461
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 5461 — Two active tablets, given daily
  Arms: ALKS 5461
Drug: Placebo — Two placebo tablets, given daily
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of ALKS 5461 when administered daily for 4 weeks to adults with Major Depressive Disorder (MDD) and inadequate response to antidepressant therapy.

DETAILED DESCRIPTION:
The study will measure efficacy using the HAM-D-17, the MADRS, and the CGI-S as well as using other scales and assessments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a major depressive episode (MDE)
* Body mass index less than or equal to 40 kg/m2
* Have been treated with an adequate dose of SSRI/SNRI during the current MDE for at least 8 weeks, with the same, adequate dose over the last 4 weeks that is expected to remain stable throughout the study
* History of inadequate response during the entire current MDE to 1 or 2 adequate antidepressant treatments, including current treatment
* Be otherwise physically healthy

Exclusion Criteria:

* Have an axis I diagnosis of delirium, dementia, amnestic or other cognitive disorder, schizophrenia or other psychotic disorder, bipolar I or II disorder, eating disorder, obsessive-compulsive disorder, panic disorder, acute stress disorder, or posttraumatic stress disorder
* Have a clinically significant current axis II diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder
* Are experiencing hallucinations, delusions, or any psychotic symptomatology in the current MDE
* Receive new onset psychotherapy within 6 weeks of screening
* Use of opioid agonists (eg, codeine, oxycodone, morphine) within 14 days before screening
* Have received electroconvulsive therapy during the current MDE
* Have attempted suicide within the past 2 years
* Have a thyroid pathology
* Have a history of a seizure disorder or of neuroleptic malignant syndrome/serotonin syndrome
* Have a positive test for human immunodeficiency virus (HIV)

Additional inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Leigh-Pemberton, MD, Study Director — Alkermes, Inc.
Locations (27):
- United States (27):
  - Alkermes Investigational Site, Tucson, Arizona
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Santa Ana, California
  - Alkermes Investigational Site, Torrance, California
  - Alkermes Investigational Site, Fort Myers, Florida
  - Alkermes Investigational Site, Lauderhill, Florida
  - Alkermes Investigational Site, Leesburg, Florida
  - Alkermes Investigational Site, North Miami, Florida
  - Alkermes Investigational Site, St. Petersburg, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Hoffman Estates, Illinois
  - Alkermes Investigational Site, Baltimore, Maryland
  - Alkermes Investigational Site, Boston, Massachusetts
  - Alkermes Investigational Site, Haverhill, Massachusetts
  - Alkermes Investigational Site, Berlin, New Jersey
  - Alkermes Investigational Site, Brooklyn, New York
  - Alkermes Investigational Site, New York, New York
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Charleston, South Carolina
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, San Antonio, Texas
  - Alkermes Investigational Site, Bellevue, Washington

REFERENCES:
- [Result] Fava M, Memisoglu A, Thase ME, Bodkin JA, Trivedi MH, de Somer M, Du Y, Leigh-Pemberton R, DiPetrillo L, Silverman B, Ehrich E. Opioid Modulation With Buprenorphine/Samidorphan as Adjunctive Treatment for Inadequate Response to Antidepressants: A Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2016 May 1;173(5):499-508. doi: 10.1176/appi.ajp.2015.15070921. Epub 2016 Feb 12. PMID 26869247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were diagnosed with major depressive disorder (MDD) and had an inadequate response to 1 or 2 adequate courses of treatment with a commercially available antidepressant therapy (ADT) during the current major depressive episode (MDE). All subjects continued ADT for the duration of the study.
Pre-assignment Details: This was a Sequential Parallel Comparison Design (SPCD) study comprised of 2 stages. In Stage 1 subjects were randomized to ALKS 5461 or placebo (2:2:9). In Stage 2 only placebo non-responders from Stage 1 were re-randomized to ALKS 5461 or placebo (1:1:1). One subject randomized to placebo did not receive study drug.
Groups:
- Placebo S1: Received placebo in Stage 1
- ALKS 5461 2mg/2mg S1: Received ALKS 5461 2mg/2mg in Stage 1
- ALKS 5461 8mg/8mg S1: Received ALKS 5461 8mg/8mg in Stage 1
- Placebo S2: Received placebo in Stage 2
- ALKS 5461 2mg/2mg S2: Received ALKS 5461 2mg/2mg in Stage 2
- ALKS 5461 8mg/8mg S2: Received ALKS 5461 8mg/8mg in Stage 2
Period: Stage 1
Arm/Group | Placebo S1 | ALKS 5461 2mg/2mg S1 | ALKS 5461 8mg/8mg S1 | Placebo S2 | ALKS 5461 2mg/2mg S2 | ALKS 5461 8mg/8mg S2
Started | 98 | 24 | 19 | 0 | 0 | 0
Completed | 90 | 18 | 13 | 0 | 0 | 0
Not Completed | 8 | 6 | 6 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 4 | 5 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Noncompliance with Study Drug | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Placebo S1 | ALKS 5461 2mg/2mg S1 | ALKS 5461 8mg/8mg S1 | Placebo S2 | ALKS 5461 2mg/2mg S2 | ALKS 5461 8mg/8mg S2
Started (Subjects in Stage 2 are a subset of those randomized to placebo in Stage 1.) | 0 | 0 | 0 | 20 | 23 | 22
Completed | 0 | 0 | 0 | 20 | 18 | 18
Not Completed | 0 | 0 | 0 | 0 | 5 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 5 | 4

BASELINE CHARACTERISTICS:
Population: All subjects randomized to Stage 1 (i.e., all subjects randomized during the study) who received ≥ dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo S1 | ALKS 5461 2mg/2mg S1 | ALKS 5461 8mg/8mg S1 | Total
Number analyzed (Participants) | 98 | 24 | 19 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (11.0) | 45.2 (10.9) | 45.8 (11.9) | 46.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 17 | 11 | 96
  Male | 30 | 7 | 8 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 23 | 9 | 6 | 38
  White | 74 | 15 | 13 | 102
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: Count of participants]
  United States | 98 | 24 | 19 | 141

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in Hamilton Rating Scale for Depression (HAM-D17) Total Score
Description: The HAM-D17 scale is a clinician-administered questionnaire comprised of 17 items used to measure the severity of MDD symptoms. Scores range from 0 (no apparent symptoms) to 50 (most severe symptoms). Individual questionnaire items include depressed mood, work and activities, insomnia (early), insomnia (middle), insomnia (late), genital symptoms, somatic symptoms (gastrointestinal), loss of weight, somatic symptoms (general), feelings of guilt, suicide, anxiety (psychic), anxiety (somatic), hypochondriasis, insight, agitation, and retardation.
Time Frame: Baseline and 4 weeks for each stage
Population: Stage 1 and Stage 2 Full Analysis Sets (FAS) consisted of subjects who were randomized and took at least 1 dose of study drug and had at least 1 postbaseline HAM-D17 assessment in the respective stage. Two subjects randomized to 8/8 in Stage 1 received 2/2. These subjects are included in the 8/8 group for efficacy analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo S1: Subjects randomized to placebo in Stage 1
- ALKS 5461 2mg/2mg S1: Subjects randomized to ALKS 5461 2mg/2mg in Stage 1
- ALKS 5461 8mg/8mg S1: Subjects randomized to ALKS 5461 8mg/8mg in Stage 1
- Placebo S2: Subjects randomized to placebo in Stage 2
- ALKS 5461 2mg/2mg S2: Subjects randomized to ALKS 5461 2mg/2mg in Stage 2
- ALKS 5461 8mg/8mg S2: Subjects randomized to ALKS 5461 8mg/8mg in Stage 2
Arm/Group | Placebo S1 | ALKS 5461 2mg/2mg S1 | ALKS 5461 8mg/8mg S1 | Placebo S2 | ALKS 5461 2mg/2mg S2 | ALKS 5461 8mg/8mg S2
Number analyzed (Participants) | 95 | 20 | 20 | 20 | 23 | 22
score on a scale | -7.1 (0.6) | -9.3 (1.5) | -6.6 (1.6) | -1.5 (1.1) | -5.2 (1.2) | -3.3 (1.1)
Statistical Analysis 1: Comparison: Placebo S1 vs ALKS 5461 2mg/2mg S1 vs Placebo S2 vs ALKS 5461 2mg/2mg S2; Analysis was conducted for each stage separately and overall efficacy was based on combined stage analysis where stage-specific estimates were combined using pre-specified weights (0.6/0.4 for Stage 1/Stage 2). Within each stage ALKS 5461 2mg/2mg was compared to placebo (i.e., ALKS 5461 2mg/2mg S1 vs Placebo S1; and ALKS 5461 2mg/2mg S2 vs Placebo S2; Test type: Superiority; p = 0.014, Mixed Models Analysis — Hypothesis tests were two-sided with an alpha of 0.5; ALKS 5461 was compared to PBO using stage-specific MMRM for change from Baseline. Model-derived estimates were combined using pre-specified weights
Statistical Analysis 2: Comparison: Placebo S1 vs ALKS 5461 8mg/8mg S1 vs Placebo S2 vs ALKS 5461 8mg/8mg S2; Analysis was conducted for each stage separately and overall efficacy was based on combined stage analysis where stage-specific estimates were combined using pre-specified weights (0.6/0.4 for Stage 1/Stage 2). Within each stage ALKS 5461 8mg/8mg was compared to placebo (i.e., ALKS 5461 8mg/8mg S1 vs Placebo S1; and ALKS 5461 8mg/8mg S2 vs Placebo S2; Test type: Superiority; p = 0.699, Mixed Models Analysis — Hypothesis tests were two-sided with an alpha of 0.05; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Proportion of Patients Who Exhibited Treatment Response (HAM-D17)
Description: The proportion of subjects demonstrating HAM-D17 treatment response, defined as a ≥ 50% reduction in HAM-D17 score from baseline to the end of the efficacy period (Week 4). The HAM-D17 is a clinician administered questionnaire comprised of 17 questions used to assess the severity of a patient's depression. Scores range from 0 (no apparent symptoms) to 50 (most severe symptoms). Individual questionnaire items include depressed mood, work and activities, insomnia (early), insomnia (middle), insomnia (late), genital symptoms, somatic symptoms (gastrointestinal), loss of weight, somatic symptoms (general), feelings of guilt, suicide, anxiety (psychic), anxiety (somatic), hypochondriasis, insight, agitation, and retardation.
Time Frame: 4 weeks for each stage
Population: Stage 1 and Stage 2 Full Analysis Sets (FAS) consisted of subjects who were randomized and took at least 1 dose of study drug and had at least 1 postbaseline HAM-D17 assessment in the respective stage.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo S1 | ALKS 5461 2mg/2mg S1 | ALKS 5461 8mg/8mg S1 | Placebo S2 | ALKS 5461 2mg/2mg S2 | ALKS 5461 8mg/8mg S2
Number analyzed (Participants) | 90 | 17 | 14 | 20 | 18 | 18
Participants
  Yes | 23 | 8 | 5 | 3 | 6 | 5
  No | 67 | 9 | 9 | 17 | 12 | 13

3. Secondary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS-10 scale is a clinician-administered questionnaire comprised of 10 items used to measure the severity of MDD symptoms. Scores range from 0 (no apparent symptoms) to 60 (most severe symptoms). Individual questionnaire items include: Apparent Sadness, Reported Sadness, Inner Tension, Reduced Sleep, Reduced Appetite, Concentration Difficulties, Lassitude, Inability to Feel, Pessimistic Thoughts, and Suicidal Thoughts.
Time Frame: 4 weeks for each stage
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo S1 | ALKS 5461 2mg/2mg S1 | ALKS 5461 8mg/8mg S1 | Placebo S2 | ALKS 5461 2mg/2mg S2 | ALKS 5461 8mg/8mg S2
Number analyzed (Participants) | 95 | 20 | 20 | 20 | 23 | 22
score on a scale | -9.6 (0.9) | -13.3 (2.2) | -11.3 (2.3) | -2.1 (1.6) | -8.8 (1.7) | -4.7 (1.7)

4. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Total Score
Description: The CGI-S is a 7-point scale that requires the clinician to assess how mentally ill the patient is at a specific point in time. Based on the scale, patients are categorized as follows: "1: normal, not at all ill"; "2: borderline mentally ill"; "3: mildly ill"; "4: moderately ill"; "5: markedly ill"; "6: severely ill"; and "7: among the most extremely ill patients."
Time Frame: 4 weeks for each stage
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo S1 | ALKS 5461 2mg/2mg S1 | ALKS 5461 8mg/8mg S1 | Placebo S2 | ALKS 5461 2mg/2mg S2 | ALKS 5461 8mg/8mg S2
Number analyzed (Participants) | 95 | 20 | 20 | 20 | 23 | 22
score on a scale | -1.0 (0.1) | -1.3 (0.2) | -1.2 (0.3) | -0.5 (0.2) | -1.1 (0.2) | -0.6 (0.2)

ADVERSE EVENTS:
Time Frame: 4 weeks for each stage
Description: The safety population includes all subjects who were randomized and received at least 1 dose of study drug. Two subjects randomized to 8/8 in Stage 1 received 2/2. These subjects are included in the 2/2 group for the safety analysis.
Groups:
- ALKS 5461 2mg/2mg S2: Received ALKS 5461 2mg/2mg in Stage 1
- ALKS 5461 8mg/8mg S2: Received ALKS 5461 8mg/8mg in Stage 1
Arm/Group | Placebo S1 | ALKS 5461 2mg/2mg S1 | ALKS 5461 8mg/8mg S1 | Placebo S2 | ALKS 5461 2mg/2mg S2 | ALKS 5461 8mg/8mg S2
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/24 | 0/19 | 0/20 | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/98 | 1/24 | 0/19 | 0/20 | 1/23 | 0/22
Other Adverse Events (participants affected / at risk) | 42/98 | 15/24 | 18/19 | 11/20 | 19/23 | 17/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo S1 (N=98) | ALKS 5461 2mg/2mg S1 (N=24) | ALKS 5461 8mg/8mg S1 (N=19) | Placebo S2 (N=20) | ALKS 5461 2mg/2mg S2 (N=23) | ALKS 5461 8mg/8mg S2 (N=22)
Multiple drug overdose intentional (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo S1 (N=98) | ALKS 5461 2mg/2mg S1 (N=24) | ALKS 5461 8mg/8mg S1 (N=19) | Placebo S2 (N=20) | ALKS 5461 2mg/2mg S2 (N=23) | ALKS 5461 8mg/8mg S2 (N=22)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 5 (6) | 9 (10) | 2 (2) | 10 (11) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (6) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (5) | 7 (7) | 1 (1) | 5 (6) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Product taste abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram RR interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 5 (5) | 4 (5) | 9 (10) | 1 (1) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 14 (19) | 1 (1) | 5 (8) | 4 (5) | 1 (2) | 5 (8)
Sedation (Nervous system disorders) | 2 (2) | 3 (4) | 5 (5) | 0 (0) | 4 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (3)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Two subjects randomized to 8/8 received 2/2 and are presented in the Participant Flow, Baseline, and AE tables by actual treatment received. For the outcome measures, subjects were analyzed by randomization treatment assignment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.